CLINICAL TRIAL: NCT05670743
Title: Pharmacokinetics of Advantage Arrest in Healthy Children 13-Months to 13-Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advantage Silver Dental Arrest, LLC (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDF PK WCGIRB-v1
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries in Children
Keywords: pharmacokinetics
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: This is a topical agent where the active ingredients are applied to the teeth and eventually swallowed and may be absorbed through the GI tract or excreted. Minimal amounts are absorbed through the oral mucosa. Serum concentrations of silver and fluoride will be be proportional to the dose of silver and fluoride administered topically to the teeth as part of Advantage Arrest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Silver diamine fluoride (Experimental): Silver diamine fluoride, 38%, topical, single application
  Interventions: Drug: 38% silver diamine fluoride

INTERVENTIONS:
Drug: 38% silver diamine fluoride — Topical application of 38% silver diamine fluoride to dental caries lesions
  Other Names: Advantage Silver Arrest

SUMMARY:
The purpose of this study is to further characterize basic pharmacokinetic (PK) parameters in healthy children to contribute to evidence for the safety of silver diamine fluoride (SDF; Advantage Arrest). Children with at least one active cavity will be treated and then have blood draws at random time points afterwards.

DETAILED DESCRIPTION:
The FDA requested additional data to evaluate the pharmacokinetics of silver diamine fluoride (SDF, Advantage Arrest) in children 13 months to 13 years old. The first request is for children under 36 months of age to be included in a study. The second request is for serum silver concentration be evaluated for a longer duration post-application to better estimate the half-life of silver and return of serum silver to baseline levels in children.

ELIGIBILITY:
Inclusion Criteria:

* At least one untreated caries lesion into the dentin
* Live within 10 miles of study site

Exclusion Criteria:

* oral mucositis
* ulcerative oral lesions
* hypersensitivity to silver or fluoride
* history of treatment with silver diamine fluoride within 3 months

Ages: 13 Months to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Fluoride Cmax | 21 days
  Maximum serum concentration of fluoride
Silver Cmax | 21 days
  Maximum serum concentration of silver
Fluoride Tmax | 21 days
  Time to maximum serum concentration of fluoride
Silver Tmax | 21 days
  Time to maximum serum concentration of silver
Area Under Curve, Fluoride | 21 days
  Area under the curve, fluoride
Area Under Curve, Silver | 21 days
  Area under the curve, silver

CONTACTS AND LOCATIONS:
Overall Officials: Travis Nelson, DDS, Principal Investigator — University of Washington
Locations (1):
- Center for Pediatric Dentistry, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No